CLINICAL TRIAL: NCT06630442
Title: Efficacy of an Educational Food Safety Intervention for Cancer Patients Receiving Treatment
Brief Title: Food Safety Educational Training Program to Improve Food Safety Knowledge and Behaviors in Cancer Patients Receiving Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sanja Ilic, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-21049; NCI-2024-06192 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (food safety educational training) (Experimental): Patients attend a food safety educational training program over 50 minutes on study.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Attend a food safety educational training program
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the impact of a food safety educational training program on food safety knowledge and behaviors in cancer patients receiving treatment. Cancer treatments, such as chemotherapy, can put patients at risk for foodborne infections and despite this risk, it has been reported that patients do not receive any food safety counseling until they are already experiencing low white blood cell counts. A food safety educational training program may help cancer patients make better choices of low-risk foods and prepare foods safely.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the efficacy of a food safety education intervention for cancer patients.

OUTLINE:

Patients attend a food safety educational training program over 50 minutes on study.

After completion of study intervention, patients are followed up at 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age
* Able to fluently read and converse in English (though it does not have to be their first language)
* All participants must be diagnosed with cancer, any stage, and be receiving some form of treatment at the aforementioned facilities
* Informed consent must be obtained from each patient prior to participation in any aspect of the study

Exclusion Criteria:

* Patients who do not meet these criteria or are not willing or are unable to give informed consent, will be excluded from this study
* Patients with prescribed dietary limitations or currently on neutropenic diet unrelated to this study will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Changes in food safety knowledge | From baseline up to 5 weeks post intervention
  Pre and post responses will be determined using score calculation and compared using analysis of variance (ANOVA).
Changes in attitudes | From baseline up to 5 weeks post intervention
  Pre and post responses will be determined using score calculation and compared using ANOVA.
Changes in risk perception | From baseline up to 5 weeks post intervention
  Pre and post responses will be determined using score calculation and compared using ANOVA.
Changes in self-efficacy | From baseline up to 5 weeks post intervention
  Pre and post responses will be determined using score calculation and compared using ANOVA.
Changes in behaviors | From baseline up to 5 weeks post intervention
  Pre and post responses will be determined using score calculation and compared using ANOVA.
Changes in food acquisition practices | From baseline up to 5 weeks post intervention
  Pre and post responses will be determined using score calculation and compared using ANOVA.
Changes in high-risk food consumption | From baseline up to 5 weeks post intervention
  Pre and post responses will be determined using score calculation and compared using ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Ilic, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT06630442/ICF_000.pdf